CLINICAL TRIAL: NCT02067156
Title: An Open-Label, Single-Arm, Phase II Study to Evaluate the Efficacy, Safety and CNS Exposure of G-202 (Mipsagargin) in Patients With Recurrent or Progressive Glioblastoma
Brief Title: Efficacy, Safety and CNS Exposure of G-202 (Mipsagargin) in Patients With Recurrent or Progressive Glioblastoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GenSpera, Inc. (Industry)
Collaborators: Food and Drug Administration (FDA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G-202-004; R01FD005077 (FDA)
Record Dates: First submitted 2014-02-16; First posted 2014-02-20 (Estimated); Results first posted 2024-05-21 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Glioblastoma Multiforme
Keywords: glioblastoma
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- G-202 (Mipsagargin) (Experimental): G-202 (Mipsagargin) administered by intravenous infusion on 3 consecutive days of a 28-day cycle
  Interventions: Drug: G-202

INTERVENTIONS:
Drug: G-202 — G-202 administered by intravenous infusion (IV, in the vein) on Days 1, 2 and 3 of each 28-day cycle until progression or development of unacceptable toxicity
  Other Names: Mipsagargin

SUMMARY:
This study will evaluate if a drug called G-202 can be safely used to treat people with glioblastoma (GBM) that has progressed or recurred. G-202 is given by intravenous infusion on three consecutive days of a 28-day cycle.

DETAILED DESCRIPTION:
Glioblastoma (GBM) comprises about 16% of all malignancies of the nervous system and over 50% of all gliomas. Standard of care for newly-diagnosed GBM is a combination of surgical debulking followed by concurrent radiotherapy and chemotherapy with temozolomide. Efforts to improve second-line therapy in GBM have met with only marginal success and there is a large unmet medical need for new therapies. G-202 (mipsagargin) is an example of prodrug chemotherapy. It is activated by Prostate Specific Membrane Antigen (PSMA), which is expressed by some cancer cells and in the blood vessels of most solid tumors, including GBM, but not by normal cells or blood vessels in normal tissue. It is believed that activation of the prodrug G-202 will allow the drug to kill cancer cells. This study will evaluate the activity, safety and CNS exposure of G-202 in participants with recurrent or progressive GBM receiving G-202 by intravenous infusion on three consecutive days of a 28-day cycle. Funding Source - FDA Office of Orphan Products Development (OOPD)

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent to participate in this study
* Histological or radiological confirmation of glioblastoma
* Recurrent or progressive GBM following at least one (1), but no more than two (2) prior regimens; one of the prior regimens must have included surgery and/or radiotherapy
* Age > 18 years
* Karnofsky Performance Status (KPS) ≥ 60%
* Life expectancy > 2 months
* Adequate hematologic, renal and hepatic function
* Adequate coagulation profile
* Not pregnant, nursing or planning to become pregnant; willing to use contraception

Exclusion Criteria:

* Deteriorating neurological symptoms, or need for increasing doses of corticosteroids or new onset of seizures
* Surgical resection or major surgery within 4 weeks or stereotactic biopsy within 1 week of first G-202 treatment
* Toxicity from prior therapy (excluding alopecia) that has not resolved to ≤ Grade 1 unless otherwise specified
* Investigational or cytotoxic therapy within 28 days or nitrosoureas within 42 days of the first treatment with G-202
* Currently requiring any type of full-dose anti-coagulation treatment, systemic administration of antibiotics or chronic administration of anti-viral agents.
* History or evidence of cardiac risk, including QTc interval on screening ECG >470 msec, left ventricular ejection fraction (LVEF) < 50%, clinically significant uncontrolled arrhythmias or arrhythmia requiring treatment with the exceptions of atrial fibrillation and paroxysmal supraventricular tachycardia, history of acute coronary syndromes within 6 months prior to the first dose of study therapy (including myocardial infarction and unstable angina, coronary artery bypass graft, angioplasty, or stenting)
* Uncontrolled cardiac or coronary artery disease
* Uncontrolled hypertension (mean systolic BP ≥ 160 mm Hg and/or mean diastolic BP ≥ 100 mm Hg on 3 determinations 5 minutes apart while on 2 anti-hypertensive agents) or hypertension requiring treatment with more than 2 anti-hypertensive agents
* Severe or uncontrolled medical disease, including uncontrolled diabetes, congestive heart failure, chronic renal disease or chronic pulmonary disease
* Severe GI bleeding within 12 weeks of treatment with G-202
* Known history of HIV, hepatitis B or hepatitis C
* Documentation of keratosis follicularis (also known as Darier or Darier-White disease)
* Requirement for chronic use of strong inhibitors or inducers of cytochrome (CYP3A4) iso-enzymes
* Known hypersensitivity to any study drug component including thapsigargin derivatives, polysorbate 20, or propylene glycol
* Any other condition, including concurrent medical condition, social circumstance or drug dependency, which in the opinion of the investigator could compromise patient safety and/or compliance with study requirements
* Another primary malignancy that has not been in remission for at least 2 years; non-melanoma skin cancer, intraepithelial carcinoma of the cervix, or prostate cancer with a current PSA ≤ 0.1 ng/mL is allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Piccioni, M.D., Ph.D., Principal Investigator — University of California, San Diego Moores Cancer Center
Locations (1):
- University of California, San Diego Moores Cancer Center, La Jolla, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | G-202 (Mipsagargin)
Started | 26
Completed | 22
Not Completed | 4
Not completed — Lost to Follow-up | 4

BASELINE CHARACTERISTICS:
Arm/Group | G-202 (Mipsagargin)
Number analyzed (Participants) | 26
Age, Continuous [Median (Full Range); unit: years] | 55 [21 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 23
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 21
  More than one race | 0
  Unknown or Not Reported | 4

OUTCOME MEASURES:

1. Primary Outcome: 6-month Progression-free Survival (PFS)
Description: Percentage of patients who received at least 2 cycles of G-202 and have not progressed or died within 6 months of beginning treatment with G-202. Progression is defined using Response Assessment in Neuro-Oncology Working Group (RANO) for high-grade glioma, as any of the following: by any of the following: 25% or greater increase in sum of the products of perpendicular diameters of enhancing lesions (compared with baseline if no decrease) on stable or increasing doses of corticosteroids; a significant increase in T2/FLAIR nonenhancing lesions on stable or increasing doses of corticosteroids compared with baseline scan or best response after initiation of therapy, not due to comorbid events; the appearance of any new lesions; clear progression of nonmeasurable lesions; or definite clinical deterioration not attributable to other causes apart from the tumor, or to decrease in corticosteroid dose.
Time Frame: 6 months
Population: response-evaluable participants
Measure: Count of Participants; unit: Participants
Arm/Group | G-202 (Mipsagargin)
Number analyzed (Participants) | 21
Participants | 1

2. Secondary Outcome: Toxicity Assessed by CTCAE v 4.03 Criteria
Description: Percentage of all analyzed patients experiencing treatment-emergent adverse events.
Time Frame: Every 2 weeks for approximately one year
Measure: Count of Participants; unit: Participants
Arm/Group | G-202 (Mipsagargin)
Number analyzed (Participants) | 26
Participants | 26

3. Secondary Outcome: Objective Tumor Response Rate
Description: Percentage of analyzed participants experiencing a complete response (CR) or partial response (PR) using RANO criteria. CR is defined as complete disappearance of all enhancing measurable and nonmeasurable disease sustained for at least 4 weeks; no new lesions; stable or improved nonenhancing (T2/FLAIR) lesions; and patient must be off corticosteroids or on physiologic replacement doses only, and stable or improved clinically. PR is defined as at least 50% decrease, compared with baseline, in the sum of products of perpendicular diameters of all measurable enhancing lesions sustained for at least 4 weeks; no progression of nonmeasurable disease; no new lesions; stable or improved nonenhancing (T2/FLAIR) lesions on same or lower dose of corticosteroids compared with baseline scan; and patient must be on a corticosteroid dose not greater than the dose at time of baseline scan and is stable or improved clinically.
Time Frame: approximately one year
Population: response-evaluable participants
Measure: Count of Participants; unit: Participants
Arm/Group | G-202 (Mipsagargin)
Number analyzed (Participants) | 21
Participants | 0

4. Secondary Outcome: Duration of PFS
Description: Duration of time from the first administration of G-202 until the first documented progression or date of death, assessed up to 12 months. Progression is defined using Response Assessment in Neuro-Oncology Working Group (RANO) for high-grade glioma, as any of the following: by any of the following: 25% or greater increase in sum of the products of perpendicular diameters of enhancing lesions (compared with baseline if no decrease) on stable or increasing doses of corticosteroids; a significant increase in T2/FLAIR nonenhancing lesions on stable or increasing doses of corticosteroids compared with baseline scan or best response after initiation of therapy, not due to comorbid events; the appearance of any new lesions; clear progression of nonmeasurable lesions; or definite clinical deterioration not attributable to other causes apart from the tumor, or to decrease in corticosteroid dose.
Time Frame: Every 4 weeks for approximately one year
Population: response-evaluable participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | G-202 (Mipsagargin)
Number analyzed (Participants) | 21
months | 1.64 [1.05 to 1.74]

5. Secondary Outcome: Overall Survival
Description: Duration of time from the first administration of G-202 until the date of death, assessed up to 12 months
Time Frame: Every 4 weeks for approximately one year
Population: response-evaluable participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | G-202 (Mipsagargin)
Number analyzed (Participants) | 21
months | 7.23 [6.08 to 17]

6. Secondary Outcome: Biomarkers in Tumor
Description: PSMA immunohistochemistry staining score on tumor tissue collected prior to start of G-202 study treatment.
  Intensity of staining was ranked on a scale of 0, 1, 2, or 3 (with 0 representing no staining and 3 representing maximum intensity): absence of staining (0), weak staining (1), medium staining (2), or strong staining (3) relative to a staining calibration curve and normalized to the image mean background intensity.
  The scoring scale does not have a title nor does it have a subscale. It is not known whether PSMA staining intensity is associated with tumor molecular phenotypes or response outcome to G-202; therefore, this was an exploratory analysis. However, the lack of objective tumor response in the trial precluded comparative analysis.
Time Frame: Within 4 weeks of receiving G-202
Population: Only 11 samples of tumor tissue collected prior to the start of study treatment (G-202) were available for immunohistochemistry. PSMA staining was not an eligibility criterion.
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | G-202 (Mipsagargin)
Number analyzed (Participants) | 11
score on a scale | 2 (1.1)

ADVERSE EVENTS:
Time Frame: one year
Arm/Group | G-202 (Mipsagargin)
All-Cause Mortality (participants affected / at risk) | 22/26
Serious Adverse Events (participants affected / at risk) | 6/26
Other Adverse Events (participants affected / at risk) | 24/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | G-202 (Mipsagargin) (N=26)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Symptomatic Vomiting (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Infusion reaction (General disorders) | 1 (1)
Creatinine increased (Investigations) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Cerebral edema (Nervous system disorders) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Vertebral dissection (Nervous system disorders) | 1 (1)
Aspiration of vomit (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure due to vomiting (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | G-202 (Mipsagargin) (N=26)
Anemia (Blood and lymphatic system disorders) | 5
Constipation (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 6 (6)
Vomiting (Gastrointestinal disorders) | 5 (5)
Fatigue (General disorders) | 3 (3)
Fever (General disorders) | 2 (2)
ALT increased (Investigations) | 9 (11)
AST increased (Investigations) | 6 (6)
Creatinine increased (Investigations) | 11 (18)
Platelet count decreased (Investigations) | 7 (9)
PTT prolonged (Investigations) | 3 (3)
White blood cells decreased (Investigations) | 3 (4)
Headache (Nervous system disorders) | 3 (4)
Seizure (Nervous system disorders) | 3 (3)
Anxiety (Psychiatric disorders) | 2 (2)
Depression (Psychiatric disorders) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 6 (6)
Hypotension (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less